CLINICAL TRIAL: NCT06969352
Title: A Multicentre, Retrospective-prospective Real-world Study: to Evaluate the Effectiveness and Safety of Vorasidenib in Patients With Isocitrate Dehydrogenase IDH1/2 Mutant Grade 2 Astrocytoma or Oligodendroglioma (VICTORIA Study)
Acronym: VICTORIA
Status: Not yet recruiting | Type: Observational
Sponsor: Servier (Tianjin) Pharmaceutical Co. LTD. (Industry)
Collaborators: Institut de Recherches Internationales Servier (I.R.I.S.) (Industry); Hainan Boyan Medical Research Co. Ltd. (Unknown); Fantastic Bioimaging Co., Ltd. (Unknown); Clinical TrialService (Guangzhou) Co.,Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: S095032-235
Record Dates: First submitted 2025-04-29; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Gliomas
MeSH Terms: conditions — Glioma | interventions — vorasidenib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- treatment group(Vorasidenib): As a real-world study, in principle, a formal visit is not mandatory. However, due to the fact that patients will be treated with new drugs and need to collect data on major efficacy, regular visits should be performed in routine clinical practice.
  Interventions: Drug: Vorasidenib
- external control group (untreated after surgery): Eligible patients are those who have MRI data available for analysis after glioma surgery (including biopsy, subtotal resection, or total resection) and at least one additional MRI scan available for analysis within the following 6 months after the index data During this period, the eligible patients who have not undergone radiotherapy or chemotherapy after resection will be included in the external control arm.

INTERVENTIONS:
Drug: Vorasidenib — Treatment group: recommended dosage in adults and paediatric patients 12 years of age and older:
  * For patients weighing at least 40 kg: 40 mg, orally, once daily.
  * For patients weighing less than 40 kg: 20 mg, orally, once daily.
  Groups: treatment group(Vorasidenib)

SUMMARY:
The goal of this Study is to evaluate the effectiveness and safety of Vorasidenib in Patients with Isocitrate dehydrogenase IDH1/2 mutant Grade 2 astrocytoma or oligodendroglioma, primary purposeis to evaluate the efficectiveness of Vorasidenib in glioma patients treated in routine clinical practice in In China, patients aged 12 and above with grade II or higher astrocytoma or oligodendroglioma with IDH1 or IDH2 mutations. The main question it aims to answer is:

if this trend is consistent with the efficacy observed in the INDIGO study, and there is not any new safety signal compared to previous research data? Researchers will compare to no treatment. Participants is not mandatory for a formal visit as it is a real-word study.However, due to the fact that patients will be treated with new drugs and need to collect data on major efficacy, regular visits should be performed in routine clinical practice.

This study is a multicenter, retrospective-and prospective real-world study, There are treatment group (Vorasidenib) and external control group (untreated after surgery).

ELIGIBILITY:
Inclusion and exclusion criteria for treatment group

Patients will be included if they meet all the following criteria:

1. Patients (female and male) aged ≥ 12 years at enrolment.
2. Patients with tissue-confirmed diagnoses of Grade 2 astrocytoma or oligodendroglioma with IDH1 or IDH2 mutation
3. Have undergone at least one prior glioma surgery (biopsy, subtotal resection, or complete resection).
4. Patients with evaluable disease based on the most recent MRI in the opinion of the treating physician. A measurable non-enhanced lesion is defined as at least one target lesion with dimensions of ≥1 cm × ≥1 cm (in two dimensions). Confirmed by a centralized IRC as minimal, non-nodular, and non-measurable enhancement.
5. The PI evaluates based on the Vorasidenib label and patients is willing plan to receive Vorasidenib
6. Be able to understand and provide written informed consent if the patient is 18 years or older, or if the patient is a minor (12 years or older and under 18 years), both the patient and their legal representative must sign the informed consent.

Patients who meet at least one of the following exclusion criteria will not be included in the study:

1. Patients who received radiotherapy, chemotherapy or other IDH inhibitor for Glioma before enrolment.
2. Patients with any contrindications to Vorasidenib

Inclusion and exclusion criteria for the external control group

Patients will be included if they meet all the following criteria:

1. Patients (female and male) aged ≥ 12 years at the index date.
2. Patients with tissue-confirmed diagnoses of Grade 2 astrocytoma or oligodendroglioma with IDH1 or IDH2 mutation
3. Have undergone at least one prior glioma surgery (biopsy, subtotal resection, or complete resection) before the index date.
4. Since the index date, the patient must have undergone at least two magnetic resonance imaging (MRI) scans with an interval of at least 6 months (±30 days), showing measurable or evaluable non-enhancing lesions. Measurable non-enhancing lesions are defined as at least one target lesion that is ≥1 cm × ≥1 cm (two-dimensional). These lesions must be centrally confirmed by the IRC (Independent Review Committee) as small, non-nodular, and nonmeasurable enhancing lesions.

6) Must have at least 6 months (±30 days) follow-up historical data since the index date without any treatment in this period.

Patients who meet at least one of the following exclusion criteria will not be included in the study:

1) Patients who received radiotherapy, chemotherapy or other IDH inhibitors for Glioma before the index date.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The data for the external control group will be retrospectively collected from West China Hospital, Beijing Tiantan Hospital, and other neurosurgical centers, as well as potentially suitable data sources (e.g., the National Brain Tumor Registry Center).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | at 6 months after the index date
  TGR at 6 months after the index date*. TGR is defined as percentage change in tumour volume from baseline.

SECONDARY OUTCOMES:
Secondary efficacy endpoint | 12 months after the index date of the last required sample patient
  TTNI, TTNI is defined as the time from enrolment to the initiation of the first subsequent anticancer therapy or death due to any causes whichever occurs earlier.
Secondary efficacy endpoint | 12 months after the index date of the last required sample patient
  rwPFS, defined as the time from enrolment to physician-documented disease progression or date of death due to any cause, whichever occurs earlier, evaluated according to the modified RANO-LGG.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - West China Lecheng Hospital Sichuan University, Qionghai, Hainan
  - West China Hospital Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No